CLINICAL TRIAL: NCT06317246
Title: Subtypes and Prognostic Factors in Erdheim-Chester Disease
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Meyer Children's Hospital IRCCS (Other)
Responsible Party: Principal Investigator, Augusto Vaglio, Associate Professor of Nephrology, Principal Investigator, Meyer Children's Hospital IRCCS
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: ECDSUB
Record Dates: First submitted 2024-02-21; First posted 2024-03-19 (Actual); Last update posted 2024-03-19 (Actual); Status verified 2024-03

CONDITIONS: Erdheim-Chester Disease
MeSH Terms: conditions — Erdheim-Chester Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Investigation of BRAF mosaicism (Experimental): The study of BRAF mosaicism will be conducted on biopsy samples from patients with ECD and other neoplasms co-occurring with the BRAFV600E mutation. The samples will be labeled with anti-Pu.1-Alexa Fluor 647 antibody (which binds to macrophages), then DNA will be extracted using FACS method and amplified using MDA (Qiagen Repli-G Single-Cell kit). Quality control will be performed using Quant-it (ThermoScientific) and Agilent 4200 TapeStation. Eligible samples will undergo digital droplet PCR (ddPCR) and sequencing. ddPCR probes for wild-type and mutant alleles will be used. Sequencing will be performed using Illumina HiSeq 2500 system
  Interventions: Genetic: Investigation of BRAF mosaicism

INTERVENTIONS:
Genetic: Investigation of BRAF mosaicism — The study of BRAF mosaicism will be conducted on biopsy samples from patients with ECD and other neoplasms co-occurring with the BRAFV600E mutation. The samples will be labeled with anti-Pu.1-Alexa Fluor 647 antibody (which binds to macrophages), then DNA will be extracted using FACS method and amplified using MDA (Qiagen Repli-G Single-Cell kit). Quality control will be performed using Quant-it (ThermoScientific) and Agilent 4200 TapeStation. Eligible samples will undergo digital droplet PCR (ddPCR) and sequencing. ddPCR probes for wild-type and mutant alleles will be used. Sequencing will be performed using Illumina HiSeq 2500 system

SUMMARY:
Erdheim-Chester Disease (ECD) is a rare form of histiocytosis characterized by the proliferation of blood cells, known as histiocytes, which infiltrate various organs and tissues, often causing irreversible damage. The causes of the pathology are still unknown. Although the disease typically affects adult individuals, cases of pediatric-onset ECD have been described. However, there is a lack of detailed information on the phenotypic characteristics of these patients, and reliable data on response to specific therapies and long-term outcomes are missing. Three patients referred to our reference center for Histiocytosis present a concomitant BRAF-mutated neoplasm. Such an association could be due to the presence of mosaicisms for the BRAF V600E mutation. Mosaicism is a biological event defined as the presence of more than one genetically dissimilar cell population in the same organism and is an increasingly studied field, both in normal and pathological conditions. If proven in ECD as well, this mechanism could contribute to providing answers to the still open questions regarding the development of this disease.

ELIGIBILITY:
Inclusion Criteria:

* Prevalent and incident patients (adults and pediatric), with histologically confirmed diagnosis of Erdheim-Chester Disease according to the latest diagnostic recommendations;
* Signing of informed consent for study participation.

Exclusion Criteria:

* Patients for whom clinical and imaging data are not available and for whom it is not possible to retrieve histological samples."

Ages: 1 Year to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 70 (Estimated)
Dates: Start 2020-09-15 (Actual); Primary Completion 2024-09-15 (Estimated); Study Completion 2024-12-15 (Estimated)

PRIMARY OUTCOMES:
Clinical characteristics of patients with Erdheim-Chester Disease | 4 years
  Evaluation of clinical characteristics in extreme subtypes of Erdheim-Chester Disease
Prognostic factors of patients with Erdheim-Chester Disease | 4 years
  Evaluation of prognostic factors in extreme subtypes of Erdheim-Chester Disease

CONTACTS AND LOCATIONS:
Locations (2):
- Italy (2):
  - Meyer Children's Hospital IRCCS, Florence, Firenze
  - AOU Parma, Parma

IPD SHARING:
Plan to Share IPD: No